CLINICAL TRIAL: NCT04827550
Title: Fatigue Levels in Fibromyalgia Syndrome and the Relationship Between Disease Activity, Kinesiophobia and Physical Activity
Brief Title: Fatigue Levels in Fibromyalgia Syndrome
Status: Completed | Type: Observational
Sponsor: Yerkoy State Hospital (Other)
Responsible Party: Principal Investigator, Başak Çiğdem Karaçay, specialist, Yerkoy State Hospital
Other Study IDs: 2017-KAEK-189_2021.03.10_18
Record Dates: First submitted 2021-03-31; First posted 2021-04-01 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Fatigue; Fibromyalgia
Keywords: Fibromyalgia Syndrome; Physical Activity; kinesiophobia
MeSH Terms: conditions — Fatigue; Fibromyalgia; Motor Activity; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STUDY GROUP: diagnosed with fibromyalgia according to the American College of Rheumatology 2010 diagnostic criteria
  Interventions: Other: STUDY
- CONTROL GROUP: 90 healthy volunteers
  Interventions: Other: STUDY

INTERVENTIONS:
Other: STUDY — Fibromyalgia Patient

SUMMARY:
Ninety (90) woman patients diagnosed with fibromyalgia according to the American College of Rheumatology 2010 diagnostic criteria and 90 healthy volunteers were included. The Fibromyalgia Impact Questionnaire (FIQ) is used to assess the patient's functionality and determine the severity of the disease. The Fatigue Severity Scale (FSS) assessed the level and severity of fatigue. The short form of the International Physical Activity Questionnaire (IPAQ-SF) used to asess physical activity levels.The kinesiophobia level was assessed by using the Tampa Scale for Kinesiophobia.

DETAILED DESCRIPTION:
Our study consists of 180 female participants aged between 18 and 65 years who applied to the physical therapy and rehabilitation outpatient clinic between April 2021 and August 2021. This case-control study was conducted according to the Declaration of Helsinki. Participants gave written voluntary consent and enrolled in this case-control study.

Ninety (90) woman patients diagnosed with fibromyalgia according to the American College of Rheumatology 2010 diagnostic criteria and 90 healthy volunteers were included. Fibromyalgia Impact Questionnaire, Tampa Kinesiophobia Scale, Fatigue Severity Scale and The short form of İnternational Physical Activity Questionnaire (IPAQ-SF) were completed. All scales were filled in face to face for the participants. In addition, demographic data (age, gender, height, weight, marital status, education level) and duration of fibromyalgia diagnosis were recorded.

Exclusion criteria for both groups; The presence of health problems that affect the level of physical activity ( Cardiac or pulmonary insufficiency, limb amputation, recent surgery history) and cognitive impairment that prevents answer questions

ELIGIBILITY:
Inclusion Criteria:

* Ninety (90) woman patients diagnosed with fibromyalgia according to the American College of Rheumatology 2010 diagnostic criteria
* Ninety (90) healthy volunteers

Exclusion Criteria:

* The presence of health problems that affect the level of physical activity ( Cardiac or pulmonary insufficiency, limb amputation, recent surgery history)
* Cognitive impairment that prevents answer questions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Our study consists of 180 female participants aged between 18 and 65 years who applied to the physical therapy and rehabilitation outpatient clinic.
Study Population: Our study consists of 180 female participants aged between 18 and 65 years who applied to the physical therapy and rehabilitation outpatient clinic between April 2021 and August 2021. This case-control study was conducted according to the Declaration of Helsinki. Participants gave written voluntary consent and enrolled in this case-control study.
  Ninety woman patients diagnosed with fibromyalgia according to the American College of Rheumatology 2010 diagnostic criteria and 90 healthy volunteers were included
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
fatigue | Baseline (0 day)
  The Fibromyalgia Impact Questionnaire (FIQ) is used to assess the patient's functionality and determine the severity of the disease. The scale consists of 10 items and each item is 10 points. Therefore, the total maximum score is 100 points. Increasing scores indicate higher disease activity and lower functional status

SECONDARY OUTCOMES:
Kinesiophobia | Baseline (0 day)
  The kinesiophobia level was assessed by using the Tampa Scale for Kinesiophobia (TSK). The TSK includes 17 item and assesses the subjective rating of kinesiophobia..Each item is scored by using a 4-point Likert-type scale, (1 point is reporting complete disagreement and 4 points is reporting complete agreement).The total points ranges between 17 and 68. Higher scores refer higher severity of kinesiophobia. Scores higher than 37 points mean high levels of kinesiophobia and scores less than or equal to 37 mean low levels of kinesiophobia

OTHER OUTCOMES:
Physical Activity Levels | Baseline (0 day)
  The short form of the International Physical Activity Questionnaire (IPAQ-SF) contains 7 questions that provide information about sitting, walking, and moderate to vigorous intensity activities. The total score includes the duration (minutes) and frequency (days) of intense activity. The sitting score (sedentary behavior level) is calculated separately. Each activity needs to be done for at least 10 minutes at a time
functionality | Baseline (0 day)
  The Fibromyalgia Impact Questionnaire (FIQ) is used to assess the patient's functionality and determine the severity of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Basak CigdemKaracay, Spesialist, Principal Investigator — Yerkoy State Hospital
Locations (1):
- Yerkoy State Hospital, Yerköy, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gencay-Can A, Can SS. Validation of the Turkish version of the fatigue severity scale in patients with fibromyalgia. Rheumatol Int. 2012 Jan;32(1):27-31. doi: 10.1007/s00296-010-1558-3. Epub 2010 Jul 24. PMID 20658235
- [Background] Bennett R. The Fibromyalgia Impact Questionnaire (FIQ): a review of its development, current version, operating characteristics and uses. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S154-62. PMID 16273800
- [Background] Burwinkle T, Robinson JP, Turk DC. Fear of movement: factor structure of the tampa scale of kinesiophobia in patients with fibromyalgia syndrome. J Pain. 2005 Jun;6(6):384-91. doi: 10.1016/j.jpain.2005.01.355. PMID 15943960
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588